CLINICAL TRIAL: NCT03665090
Title: A Three-year Community-based Study in Diabetes: The Shanghai Cohort Study of Diabetic Eye Disease
Brief Title: Shanghai Cohort Study of Diabetic Eye Disease
Acronym: SCODE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Principal Investigator, Jiannan Huang, Principal Investigator, Shanghai Eye Disease Prevention and Treatment Center
Other Study IDs: YFZX2018007
Record Dates: First submitted 2018-08-30; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Macular Edema of Both Eyes (Diagnosis); Diabetic Retinopathy Visually Threatening
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and Blood Sample Collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Diabetic eye disease screening — Community-based, prospective cohort study from three consecutive years (2016 to 2018) to determine the prevalence and impact of diabetic eye disease, especially diabetic retinopathy (DR), in adults with diabetes living in Shanghai.

SUMMARY:
To describe the design, methodology and baseline characteristics of the Shanghai Cohort study of Diabetic Eye disease (SCODE) study, a community-based study to determine the prevalence and impact of diabetic eye disease, especially diabetic retinopathy (DR), in adults with diabetes living in Shanghai.

DETAILED DESCRIPTION:
The Shanghai Cohort study of Diabetic Eye disease (SCODE) was a three-year community-based study to carry out a regular ocular health screening and epidemiological analysis for diabetic eye disease in the approximately 8,000 middle-aged and elderly people with diabetes in Shanghai. Through this study, we hope to understand the prevalence, epidemic trend and the features of risk factors distribution on diabetic eye disease, especially on DR.

Meanwhile, our aims also included estimating the ocular fundus changes and visual impairment associated with different grade of DR. Furthermore, the aim of the present study was to investigate the association between serum and urine biochemical parameters and DR.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes aged 35 years and above; under archives management; residing in Shanghai.

Exclusion Criteria:

* All the study participants have difficulties of mobility or communication.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the enrolled participants got a yearly examination of diabetic eye disease for three years. Considering that the prevalence of DR gradually increases with age, the target population included adults with diabetes aged 35 years and above under archives management, residing in Shanghai. And the study participants were expected to be freely mobile, clear-thinking, and capable of cooperating to complete the ophthalmic examinations.
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence rate of diabetic eye disease | December 31, 2018
  SCODE was performed to evaluate the prevalence and rate of new cases of diabetic eye disease, especially DR, in a three-year community-based cohort study for the people with diabetes, and to identify the associated factors related with diabetic eye disease.

SECONDARY OUTCOMES:
Grading of DR | December 31, 2018
  Fundus changes were evaluated on non-mydriatic fundus photography and slit-lamp examination. Meanwhile, we will estimate the fundus changes associated with different grade of DR.
Retinal and choroidal thickness | December 31, 2018
  Retinal and choroidal thickness were evaluated on SS-OCT.
Retinal blood flow | December 31, 2018
  Retinal blood flow were evaluated on SD-OCTA.
Blood biochemistry indexes | December 31, 2018
  Blood samples were used for testing, including glucose, glycosylated hemoglobin (HbA1C), serum lipids, etc.
Urine biochemistry indexes | December 31, 2018
  Urine samples were used for testing urine albumin and creatinine.
Visual impairment | December 31, 2018
  Main Cause of visual impairment were determined by two ophthalmologists based on the ophthalmic examinations and reported history. Moreover, we will evaluate the association between the visual impairment and different grade of DR.

IPD SHARING:
Plan to Share IPD: Yes
Identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available with in one year of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Xiang Z, Lin S, Xu Y, Lu L, Shi Y, Wang Y, Yang Q, Ling S, Zhou D, Qin X, Cheng M, Zou H, Ma Y. The effects of physical activity on diabetic retinopathy in type 2 diabetes using automated vascular analysis: a cohort study. J Glob Health. 2025 Dec 5;15:04319. doi: 10.7189/jogh.15.04319. PMID 41343177